CLINICAL TRIAL: NCT03749265
Title: Rate Of Residual Clubfoot Deformity With Correlation To Absence Of Peroneus Tertius Muscle: A Prospective Study
Brief Title: Rate Of Residual Clubfoot Deformity With Correlation To Absence Of Peroneus Tertius Muscle
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Eytan Dujovny, Senior doctor in orthopedics department, HaEmek Medical Center, Israel
Other Study IDs: EMC-0010-18
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Clubfoot
Keywords: Peroneus Tertius Muscle
MeSH Terms: conditions — Clubfoot | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound test — patients need to undergo an ultrasound test for detecting the presence or abscence of peroneus tertius tendon

SUMMARY:
Rate Of Residual Clubfoot Deformity With Correlation To Absence Of Peroneus Tertius Muscle , A Prospective Study.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 5-17 years , which were treated with the Ponseti technique for Clubfoot in HaEmek medical center, and have sufficient data/follow-up about them in medical records /

Exclusion Criteria:

* patients aged< 5 years
* Neurological Clubfoot
* patients with insufficient data in medical records
* clubfoot caused by arthrogryposis , connective tissue diseases and congenital fibular hemimelia

Ages: 5 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 5-17 years , which were treated with the Ponseti technique for Clubfoot in HaEmek medical center, and have sufficient data/follow-up about them in medical records
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Presence or Absence of peroneus tertius | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Eytan Dujovni, senior, Principal Investigator — haemek medical center

IPD SHARING:
Plan to Share IPD: No